CLINICAL TRIAL: NCT02475720
Title: Survey on the Treatment Reality of Patients With EGFR Mutation-positive Non-small Cell Lung Cancer
Brief Title: Survey on the Treatment Reality of Patients With Epidermal Growth Factor Receptor (EGFR) Mutation-positive Non-small Cell Lung Cancer(NSCLC)
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D7913R00015
Record Dates: First submitted 2015-06-12; First posted 2015-06-19 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
According to the recent report using EGFR tyrosine kinase inhibitors (EGFR-TKI), there is all over survival of the EGFR gene mutation-positive NSCLC in a tendency to extension. However, the real situation and the reason are not clarified.This observational study collects the data of EGFR gene mutation-positive NSCLC approximately 2,000 from the medical record of approximately 20 facilities in Japan and observes the treatment reality of EGFR gene mutation-positive NSCLC.

DETAILED DESCRIPTION:
Study Site(s), number of subjects and countries planned Approximately 2000, Advanced Non Small Cell Lung cancer (aNSCLC) patients who fulfil the inclusion/exclusion criteria will be recruited by 10 to 20 investigational sites in Japan.

Total planned Study period Estimated date of first subject in June , 2015 Estimated date of last subject in November , 2015 Estimated date of data base lock December, 2015 Estimated date of first subject in for investigation of survival January, 2016 Estimated date of last subject in for investigation of survival March, 2016 Estimated date of data base lock for investigation of survival March, 2016

Medicinal Products (type, dose, mode of administration) and concomitant medication Not applicable Study Rationale As its benefits in EGFR mutation-positive patients have been reported, EGFR-TKI is now recommended by guidelines as standard first-line therapy for EGFR mutation-positive patients. Back then when concomitant use of platinum medication and 3rd-generation cytocidal drug was the standard therapy, treatment was of very poor prognosis, 8 to 10 months in terms of median overall survival, and a 1-year survival rate of 30% to 35%. Then, gefitinib was approved in July 2002. Takano et al. reported that survival among patients with EGFR mutation-positive non-small cell lung cancer has been getting longer after approval of gefitinib. The overall survival of patients with EGFR mutation-positive non-small cell lung cancer was 27.7 months in gefitinib group of Study North East Japan (NEJ) 002 reported by Inoue et al. in 2013, 34.8 months in gefitinib group of Study West Japan Oncology Group (WJOG) 3405 reported by Yoshioka et al. in 2014, 36.3 months in patients receiving erlotinib in Study Japan Oncology (JO) 22903 reported by Katakami et al. in 2014, and 46.9 months in afatinib group and 35.8 months in chemotherapy group of the Japanese subset in Study Lux-Lung3 reported by Kato. According to recent reports, overall survival tends to be prolonging, but the actual situation and the reason for such tendency has not been revealed.

Thus, we planned the present study, which clarify the prognosis, patient characteristics and treatment regimen of the patients with EGFR mutation positive NSCLC to provide useful information in order to promote individualized therapy for the patients with EGFR mutation positive NSCLC.

Study Objectives The primary objective of this study is intended to reveal the characteristics of and reality of the treatment and survival among patients with EGFR mutation-positive advanced/recurrent non-small cell lung cancer. The primary objective, secondary objective and exploratory objective of the study are as follows.

Primary objective of the study is:

- To estimate overall survival of the patients

Secondary objectives of the study are:

* To estimate overall survival by patient background
* To estimate overall survival by treatment sequence
* To calculate treatment time and exposure rate by treatment category (Sum of all treatment time for the patients with each treatment category/Sum of all treatment time for all patients)
* To estimate efficacy of Gefitinib treatment

Exploratory objectives of the study are:

* To explore any factors for which an impact on prognosis among patients
* To explore the relationship between treatment sequences and prognosis among patients Study Design This is a domestic, multicenter, retrospective and non-interventional diagnostic study. The data for the subjects with EGFR mutation-positive advanced/recurrent NSCLC will be collected at least 2000 cases from 10 to 20 sites.

Target subject population The patients with EGFR mutation-positive advanced/recurrent non-small cell lung cancer.

Survey items

1. Patient characteristics i) Date of NSCLC diagnosis ii) Gender (Male/Female) iii) Age at the time of diagnosis iv) Histological type (adenocarcinoma/squamous cell carcinoma/large cell carcinoma/others) v) Clinical staging at the initial diagnosis (IIIB /IV, post-operative relapse) vi) Performance Status(PS) (0/1/2/3/4), *Eastern Cooperative Oncology Group(ECOG) Performance Status vii) Smoking history (Yes/No) viii) Smoking exposure(pack year) xi) Type of EGFR mutation x) Distant metastasis organ
2. Survival status as of the end of December 2014, date of death or date of last follow-up of survival. A death with disease progression should be noted in Electronic Data Capture (EDC), but not be reported as serious adverse events unless the disease progression is greater than anticipated in the natural course of the disease. Survival status as of the end of December 2015, date of last follow-up of survival will be investigated.
3. NSCLC treatment provided for each line of treatment Name of drug category ( (i) EGFR-TKI (Gefitinib or other), (ii) Singlet Chemo, (iii) Doublet Chemo, (iv) EGFR-TKI+Chemo) The date treatment was commenced The date of last dose PS at the commencement of therapy given for each line of treatment *ECOG Performance Status Best response for each therapy (based on clinical evaluation) Total numbers of treatment cycle conducted (chemotherapy) The date on which Progressive Desease (PD) was confirmed

   * The date on which PD was evaluated by Response Evaluation Criteria in Solid Tumors（RECIST） (ver1.1)
   * The date on clinical PD is defined as disease progression met one of the any conditions below (Modified from original source)

     * Occurrence of clinical symptom by Disease Progression
     * Decreasing PS by Disease Progression
     * Occurrence of threatening condition in main organ (lymphangiosis carcinomatosa, bone marrow metastasis, carcinomatous meningitis, liver metastasis with liver disorder, etc)
     * Aggravation of the lesion in multiple organ with or without the symptom

Source :Paul A. Bunn EGFR and Anaplastic Lymphoma Kinase (ALK) TKI Therapy in Advanced NSCLC: Molecular Basis and When and Why to Stop or Change. Molecular Testing for Non-Small Cell Lung Cancer: Critical Questions, 2012 Chicago Multidisciplinary Symposium in Thoracic Oncology

Statistical methods Data collected will be analyzed using a method appropriate for the descriptive statistics in epidemiological studies. Patient characteristics will be summarized using descriptive statistics. Statistical Analysis Plan (SAP) will be prepared before database lock.

ELIGIBILITY:
Inclusion Criteria:

* 1. EGFR mutation-positive progress recurrent non-small cell lung cancer subject.
* 2. Subjects who commenced on first-line treatment between January, 2008 and December 2012.

Exclusion Criteria:

* 1. Patients has a treatment history with the drug which was not approved for marketing authorization as of 31th December , 2014
* 2. Person who were planning and/or getting involved in this survey. (applies to both AstraZeneca staff and/or staff at the study site)
* 3. Previous enrolment in the present study.
* 4. Patient was not evaluated to be appropriate for study enrolment by the investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 2000, Advanced Non Small Cell Lung cancer (aNSCLC) patients who fulfil the inclusion/exclusion criteria will be recruited by 10 to 20 investigational sites in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2015-06-19 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Overall survival of the patients. | Up to 3 monthes. Data will be collected retrospectively from medical records.Survival status as of the end of December 2014, date of death or date of last follow-up of survival.

SECONDARY OUTCOMES:
Overall survival by patient background | Up to 3 monthes. Data will be collected retrospectively from medical records.
Overall survival by treatment sequence | Up to 3 monthes. Data will be collected retrospectively from medical records.
Treatment time by treatment category | Up to 3 monthes. Data will be collected retrospectively from medical records.
Time to Treatment Failure (TTF) of Gefitinib treatment | Up to 3 monthes. Data will be collected retrospectively from medical records.

CONTACTS AND LOCATIONS:
Locations (1):
- Izumi Municipal Hospital, Izumi, Osaka, Japan

REFERENCES:
- See also: D7913R00015_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3912&filename=D7913R00015_redacted_CSR_Synopsis_FIX.pdf